CLINICAL TRIAL: NCT02523573
Title: High Flow Nasal Oxygen for Bronchoscopy With Bronchoalveolar Lavage in Acute Respiratory Failure Patients: the OptiBAL Study.
Brief Title: Study of High Flow Nasal Cannula Oxygen for Bronchoscopy With Bronchoalveolar Lavage in ICU Patients
Acronym: Optibal
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Collaborators: Tenon Hospital, Paris (Other); Henri Mondor University Hospital (Other); Hopital Antoine Beclere (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor of Intensive Care Medicine, Assistant Head of Medico-Surgical ICU, Hôpital Louis Mourier
Other Study IDs: HLM_JDR4
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: Adult ARF ICU patients needing BAL with HFNC
  Interventions: Procedure: Adult ARF ICU patients needing BAL with HFNC

INTERVENTIONS:
Procedure: Adult ARF ICU patients needing BAL with HFNC — bronchoalveolar lavage is performed in spontaneously breathing patients under high flow nasal cannula oxygen

SUMMARY:
Bronchoscopy with bronchoalveolar lavage (BAL) is at risk for worsening hypoxemia in patients with acute respiratory failure (ARF). High-flow nasal cannula oxygen (HFNC) improves hypoxemia in ARF patients . We investigated its efficacy and tolerance in intensive care unit patients admitted for ARF requiring BAL.

DETAILED DESCRIPTION:
Prospective, observational, multicenter study in ARF patients (minimal pulse oximetry -SpO2- of 92% with an minimal oxygen flow of 6 L/min , respiratory rate > 25/min (20/min if use of accessory respiratory muscles) with a compatible etiology. Primary outcome measure is increase in ventilatory support (non-invasive positive pressure ventilation (NPPV) or endotracheal intubation (ETI)) within the first 24h following BAL.

ELIGIBILITY:
Inclusion Criteria:

* presence of acute respiratory failure: defined as respiratory rate greater than 25/min, (or greater than 20/min if use of accessory respiratory muscles was present), in patients requiring oxygen greater than or equal to 6 L/min to obtain a pulse oximetry greater than 92%
* need for bronchoalveolar lavage (decision to perform BAL was left at the physician's discretion)

Exclusion Criteria:

* at least one contraindication to the bronchoscopy with BAL: acute coronary syndrome within 6 weeks; neurologic failure; thrombocytopenia less than 30 000/mm3; respiratory acidosis with a pH lower than 7.30 or hypercapnia higher than 60 mmHg; pneumothorax undrained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Intensive Care Unit, with acute hypoxemic respiratory failure requiring bronchoalveolar lavage
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
increase in ventilatory support | 24h
  increase in ventilatory support (non-invasive positive pressure ventilation (NPPV) or endotracheal intubation (ETI)) within the first 24h following BAL

SECONDARY OUTCOMES:
Immediate tolerance of bronchoscopy and BAL | 12h
  Vital signs, dyspnea score
Operator's satisfaction | 15min
  Physician performing the BAL procedure rated their comfort with HFNC from 0 to 10

OTHER OUTCOMES:
Diagnosis yield of BAL | 48h

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice La Combe, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Hopital Antoine Béclère, Clamart
  - Louis Mourier Hospital, Colombes
  - Hopital Henri Mondor, Créteil
  - Hôpital Tenon, Paris

REFERENCES:
- [Background] Messika J, Ben Ahmed K, Gaudry S, Miguel-Montanes R, Rafat C, Sztrymf B, Dreyfuss D, Ricard JD. Use of High-Flow Nasal Cannula Oxygen Therapy in Subjects With ARDS: A 1-Year Observational Study. Respir Care. 2015 Feb;60(2):162-9. doi: 10.4187/respcare.03423. Epub 2014 Nov 4. PMID 25371400
- [Background] Ricard JD. High flow nasal oxygen in acute respiratory failure. Minerva Anestesiol. 2012 Jul;78(7):836-41. Epub 2012 Apr 24. PMID 22531566
- [Background] Sztrymf B, Messika J, Bertrand F, Hurel D, Leon R, Dreyfuss D, Ricard JD. Beneficial effects of humidified high flow nasal oxygen in critical care patients: a prospective pilot study. Intensive Care Med. 2011 Nov;37(11):1780-6. doi: 10.1007/s00134-011-2354-6. Epub 2011 Sep 27. PMID 21946925
- [Result] Simon M, Braune S, Frings D, Wiontzek AK, Klose H, Kluge S. High-flow nasal cannula oxygen versus non-invasive ventilation in patients with acute hypoxaemic respiratory failure undergoing flexible bronchoscopy--a prospective randomised trial. Crit Care. 2014 Dec 22;18(6):712. doi: 10.1186/s13054-014-0712-9. PMID 25529351
- [Result] Lucangelo U, Vassallo FG, Marras E, Ferluga M, Beziza E, Comuzzi L, Berlot G, Zin WA. High-flow nasal interface improves oxygenation in patients undergoing bronchoscopy. Crit Care Res Pract. 2012;2012:506382. doi: 10.1155/2012/506382. Epub 2012 May 20. PMID 22666567
- [Result] Maitre B, Jaber S, Maggiore SM, Bergot E, Richard JC, Bakthiari H, Housset B, Boussignac G, Brochard L. Continuous positive airway pressure during fiberoptic bronchoscopy in hypoxemic patients. A randomized double-blind study using a new device. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1063-7. doi: 10.1164/ajrccm.162.3.9910117. PMID 10988131
- [Derived] La Combe B, Messika J, Labbe V, Razazi K, Maitre B, Sztrymf B, Dreyfuss D, Fartoukh M, Ricard JD. High-flow nasal oxygen for bronchoalveolar lavage in acute respiratory failure patients. Eur Respir J. 2016 Apr;47(4):1283-6. doi: 10.1183/13993003.01883-2015. Epub 2016 Feb 11. No abstract available. PMID 26869676